CLINICAL TRIAL: NCT04529304
Title: EEG-based Depth of Anesthesia-monitoring During General Anesthesia - Effects on Time to Wake-up and Post-operative Cognition
Brief Title: EEG-based Depth of Anesthesia-monitoring, Effects on Dosage and Cognition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Luis George Romundstad, Principal Investigator, Medical Doctor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2019/32173
Record Dates: First submitted 2020-03-13; First posted 2020-08-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Complications; Delayed Emergence From Anesthesia; Cognitive Dysfunction
Keywords: Depth of Anesthesia Monitoring; Post operative cognitive dysfunction (POCD)
MeSH Terms: conditions — Postoperative Complications; Delayed Emergence from Anesthesia; Cognitive Dysfunction | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Two groups with 50 participants in each group. We want to compare one group with visible EEG-monitor with a group where the EEG monitor is invisible to the anesthetic team.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient is blinded to intervention. Outcome assessoring done by patient/IPAD-solution from CANTAB, patient status assessed by blinded care-provider (nurse)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual EEG (Experimental): Individual dosing of anesthetic medications based on EEG AND other standardized clinical observations (BP, HR)
  Interventions: Device: Bilateral Bispectral Index and EEG
- Blinded EEG (Experimental): Individual dosing of anesthetic medications based on standardized clinical observations (BP, HR).
  Interventions: Device: Bilateral Bispectral Index and EEG

INTERVENTIONS:
Device: Bilateral Bispectral Index and EEG — raw-EEG and spectrographic EEG-visualization based on the Medtronic Device "Bilateral BiSpectral Index"

SUMMARY:
Depth of anesthesia-monitoring based on EEG changes demands knowledge about the effects of the different anesthetic medications on EEG waveforms. The investigators want to investigate the use of the raw-EEG waveform in addition to indexes (BIS) and EEG spectrogram analyses for depth of anesthesia monitoring. The investigators hypothesize that with the use of this monitoring, anaesthesia providers will be able to better individualize the dosage of anesthetic drugs, and that this will reduce the total consumption of anesthetic medication , thus reducing time to wake-up after surgery. Some studies have indicated that too deep anesthesia, confirmed by "burst-suppression" or isoelectric-EEG , is associated with increased postoperative cognitive dysfunction (POCD). The investigators will therefore assess the patients with the Cambridge Neuropsychological Test Automated Battery tests in mild cognitive impairment (CANTAB-MCI) cognitive function assessment tool.

DETAILED DESCRIPTION:
It has been over 80 years since Gibbs et al showed how the electroencephalogram (EEG) systematically changed in concurrence with increasing doses of hypnotic drugs such as penthobarbital and Ether. The study concluded that "Electroencephalography may therefore be of value in controlling depth of anesthesia and sedation". In spite of a solid documentation of the systematic connection between dosing of anesthetic drugs, EEG-patterns and level of sedation/anesthesia , EEG-based DoA has not become a part of standard of care in anesthetic management. There is abundant evidence of how different anesthetic drugs leads to characteristic fluctuations in human brain electrical activity, relating to depth of anesthesia, anesthetic drug of choice, and age . These anesthetic induced fluctuations are readily visible as changes in the patients EEG.

Anesthetic drugs are usually administered in pharmacological models based on a population taking into account their age, weight and height. However, there is a significant difference in how patients respond to these models. In adults there is evidence that the doses needed to achieve consciousness varies with a factor of 2 above and below suggested doses. In under-dosing of anesthetics there is a risk of peroperative awareness . On the other hand there is also evidence that overdosing of anesthetics has harmful effects; children receiving more than 4% Sevoflurane can demonstrate epileptiform activity , and adults overdosing into "burst suppression" during anesthesia has a higher risk of postoperative delirium (POD) and increased occurrence of postoperative cognitive dysfunction (POCD) .

Bispectral Index (BIS) is an algorithm developed by Aspect Medical Systems in 1994, which is based on weighted sums of EEG subparameters to present an index from 0 to 100 for depth of anesthesia, where 100 is wide awake, and 0 is an isoelectric EEG. The BIS target for a deep enough anesthesia is set to be between 40 and 60. The BIS number is often in concurrence with other clinical observations related to anesthetic depth, however there is also an experience of divergence. BIS and other EEG-based indices are programmed from adult cohorts, and cannot be directly trusted in children, or the elderly . There is also an incapability in these preprogrammed indices (BIS and other) to integrate how specific anesthetic drugs affect the EEG, and thenceforth the BIS value. An example of this is how the drug Ketamine induces a specific gamma-frequency in the EEG, which the BIS-index translate as a lighter anesthesia, even though the drug is administered "on top of" an already deep level of anesthesia.

ELIGIBILITY:
Inclusion Criteria

.

Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Participant must be above the age of 18 years , at the time of signing the informed consent.

   Sex
2. Male and/or female

   Informed Consent
3. Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol

   Exclusion Criteria

   Participants are excluded from the study if any of the following criteria apply:
4. Psychiatric disorders
5. Pregnancy
6. Breast feeding
7. Using antiepileptic drugs.
8. Central neurological disease
9. Unable to complete baseline CANTAB-test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
EEG-based Depth of anesthesia-monitoring and dosage of anesthetic medications | 24 hours
  Summarizing the total amount of anesthetic drugs used, mg/kg/hr
EEG-based Depth of anesthesia-monitoring and dosage of vasopressor medications during anesthesia | 24 hours
  Summarizing the total amount of vasopressor drugs used, micg/kg/min
EEG-based Depth of anesthesia-monitoring and time to wake-up after surgery | 24 hours
  Time from the end of intravenous infusion of anesthetic - to motoric and verbal response.
Evaluation of cognitive function using CANTAB-MCI | 1 day preoperatively to 24 hours after wake-up
  Baseline assessment 1 day preoperatively, assessment 2-3 hours after wake-up, and 24 hours after wake-up using CANTAB-MCI

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Romundstad, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data storage and management will follow GCP and GDPR requirements. Data sharing after end of study will follow the current data sharing policy at Oslo University Hospital. Data set can be made available for journal peer review process.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After end of study, 2025, and 5 years.
Access Criteria: Access through application to study contactpersons.

REFERENCES:
- [Background] Gibbs FA, Gibbs LE, Lennox WG. Effects on the electroencephalogram of certain drugs which influence nervous activity. Arch Intern Med. 1937;60:154-66
- [Background] KIERSEY DK, BICKFORD RG, FAULCONER A Jr. Electro-encephalographic patterns produced by thiopental sodium during surgical operations; description and classification. Br J Anaesth. 1951 Jul;23(3):141-52. doi: 10.1093/bja/23.3.141. No abstract available. PMID 14848401
- [Background] Tinker JH, Sharbrough FW, Michenfelder JD. Anterior shift of the dominant EEG rhytham during anesthesia in the Java monkey: correlation with anesthetic potency. Anesthesiology. 1977 Apr;46(4):252-9. doi: 10.1097/00000542-197704000-00005. PMID 402870
- [Background] John ER, Prichep LS, Kox W, Valdes-Sosa P, Bosch-Bayard J, Aubert E, Tom M, di Michele F, Gugino LD. Invariant reversible QEEG effects of anesthetics. Conscious Cogn. 2001 Jun;10(2):165-83. doi: 10.1006/ccog.2001.0507. PMID 11414713
- [Background] Gugino LD, Chabot RJ, Prichep LS, John ER, Formanek V, Aglio LS. Quantitative EEG changes associated with loss and return of consciousness in healthy adult volunteers anaesthetized with propofol or sevoflurane. Br J Anaesth. 2001 Sep;87(3):421-8. doi: 10.1093/bja/87.3.421. PMID 11517126
- [Background] Feshchenko VA, Veselis RA, Reinsel RA. Propofol-induced alpha rhythm. Neuropsychobiology. 2004;50(3):257-66. doi: 10.1159/000079981. PMID 15365226
- [Background] Cimenser A, Purdon PL, Pierce ET, Walsh JL, Salazar-Gomez AF, Harrell PG, Tavares-Stoeckel C, Habeeb K, Brown EN. Tracking brain states under general anesthesia by using global coherence analysis. Proc Natl Acad Sci U S A. 2011 May 24;108(21):8832-7. doi: 10.1073/pnas.1017041108. Epub 2011 May 9. PMID 21555565
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Ching S, Cimenser A, Purdon PL, Brown EN, Kopell NJ. Thalamocortical model for a propofol-induced alpha-rhythm associated with loss of consciousness. Proc Natl Acad Sci U S A. 2010 Dec 28;107(52):22665-70. doi: 10.1073/pnas.1017069108. Epub 2010 Dec 13. PMID 21149695
- [Background] Supp GG, Siegel M, Hipp JF, Engel AK. Cortical hypersynchrony predicts breakdown of sensory processing during loss of consciousness. Curr Biol. 2011 Dec 6;21(23):1988-93. doi: 10.1016/j.cub.2011.10.017. Epub 2011 Nov 17. PMID 22100063
- [Background] Chauvette S, Crochet S, Volgushev M, Timofeev I. Properties of slow oscillation during slow-wave sleep and anesthesia in cats. J Neurosci. 2011 Oct 19;31(42):14998-5008. doi: 10.1523/JNEUROSCI.2339-11.2011. PMID 22016533
- [Background] Lewis LD, Weiner VS, Mukamel EA, Donoghue JA, Eskandar EN, Madsen JR, Anderson WS, Hochberg LR, Cash SS, Brown EN, Purdon PL. Rapid fragmentation of neuronal networks at the onset of propofol-induced unconsciousness. Proc Natl Acad Sci U S A. 2012 Dec 4;109(49):E3377-86. doi: 10.1073/pnas.1210907109. Epub 2012 Nov 5. PMID 23129622
- [Background] Li D, Voss LJ, Sleigh JW, Li X. Effects of volatile anesthetic agents on cerebral cortical synchronization in sheep. Anesthesiology. 2013 Jul;119(1):81-8. doi: 10.1097/ALN.0b013e31828e894f. PMID 23508217
- [Background] Wang K, Steyn-Ross ML, Steyn-Ross DA, Wilson MT, Sleigh JW. EEG slow-wave coherence changes in propofol-induced general anesthesia: experiment and theory. Front Syst Neurosci. 2014 Oct 29;8:215. doi: 10.3389/fnsys.2014.00215. eCollection 2014. PMID 25400558
- [Background] Vizuete JA, Pillay S, Ropella KM, Hudetz AG. Graded defragmentation of cortical neuronal firing during recovery of consciousness in rats. Neuroscience. 2014 Sep 5;275:340-51. doi: 10.1016/j.neuroscience.2014.06.018. Epub 2014 Jun 18. PMID 24952333
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Lee JM, Akeju O, Terzakis K, Pavone KJ, Deng H, Houle TT, Firth PG, Shank ES, Brown EN, Purdon PL. A Prospective Study of Age-dependent Changes in Propofol-induced Electroencephalogram Oscillations in Children. Anesthesiology. 2017 Aug;127(2):293-306. doi: 10.1097/ALN.0000000000001717. PMID 28657957
- [Background] Iwakiri H, Nishihara N, Nagata O, Matsukawa T, Ozaki M, Sessler DI. Individual effect-site concentrations of propofol are similar at loss of consciousness and at awakening. Anesth Analg. 2005 Jan;100(1):107-110. doi: 10.1213/01.ANE.0000139358.15909.EA. PMID 15616062
- [Background] Avidan MS, Jacobsohn E, Glick D, Burnside BA, Zhang L, Villafranca A, Karl L, Kamal S, Torres B, O'Connor M, Evers AS, Gradwohl S, Lin N, Palanca BJ, Mashour GA; BAG-RECALL Research Group. Prevention of intraoperative awareness in a high-risk surgical population. N Engl J Med. 2011 Aug 18;365(7):591-600. doi: 10.1056/NEJMoa1100403. PMID 21848460
- [Background] Palanca BJ, Mashour GA, Avidan MS. Processed electroencephalogram in depth of anesthesia monitoring. Curr Opin Anaesthesiol. 2009 Oct;22(5):553-9. doi: 10.1097/ACO.0b013e3283304032. PMID 19652597
- [Background] Constant I, Sabourdin N. The EEG signal: a window on the cortical brain activity. Paediatr Anaesth. 2012 Jun;22(6):539-52. doi: 10.1111/j.1460-9592.2012.03883.x. PMID 22594406
- [Background] Gibert S, Sabourdin N, Louvet N, Moutard ML, Piat V, Guye ML, Rigouzzo A, Constant I. Epileptogenic effect of sevoflurane: determination of the minimal alveolar concentration of sevoflurane associated with major epileptoid signs in children. Anesthesiology. 2012 Dec;117(6):1253-61. doi: 10.1097/ALN.0b013e318273e272. PMID 23103557
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189
- [Background] Samarkandi AH. The bispectral index system in pediatrics--is it related to the end-tidal concentration of inhalation anesthetics? Middle East J Anaesthesiol. 2006 Feb;18(4):769-78. PMID 16749571
- [Background] Tirel O, Wodey E, Harris R, Bansard JY, Ecoffey C, Senhadji L. Variation of bispectral index under TIVA with propofol in a paediatric population. Br J Anaesth. 2008 Jan;100(1):82-7. doi: 10.1093/bja/aem339. PMID 18070785
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Hajat Z, Ahmad N, Andrzejowski J. The role and limitations of EEG-based depth of anaesthesia monitoring in theatres and intensive care. Anaesthesia. 2017 Jan;72 Suppl 1:38-47. doi: 10.1111/anae.13739. PMID 28044337
- [Background] Chhabra A, Subramaniam R, Srivastava A, Prabhakar H, Kalaivani M, Paranjape S. Spectral entropy monitoring for adults and children undergoing general anaesthesia. Cochrane Database Syst Rev. 2016 Mar 14;3(3):CD010135. doi: 10.1002/14651858.CD010135.pub2. PMID 26976247
- [Background] Juel, Bjørn Erik; Romundstad, Luis Georg; Kolstad, Frode; Storm, Johan Frederik; Larsson, Pål Gunnar. Changes in EEG captured by Directed Transfer Function is sufficient to accurately classify the state of wakefulness in patients undergoing sevoflurane anesthesia in accordance with the clinician's judgement. FENS; 2018
- [Background] Juel, Bjørn Erik; Kusztor, Aniko; Nilsen, Andre Sevenius; Farnes, Nadine; Larsson, Pål Gunnar; Romundstad, Luis Georg; Storm, Johan Frederik. Changes in electrophysiological markers of consciousness in response to various anesthetics. Nordic Neuroscience; 2017
- [Background] Juel BE, Romundstad L, Kolstad F, Storm JF, Larsson PG. Distinguishing Anesthetized from Awake State in Patients: A New Approach Using One Second Segments of Raw EEG. Front Hum Neurosci. 2018 Feb 20;12:40. doi: 10.3389/fnhum.2018.00040. eCollection 2018. PMID 29515381
- [Background] Nadine Farnes, Bjørn Erik Juel, André Sevenius Nilsen, Luis Romundstad, Johan Fredrik Storm Increased signal diversity/complexity of spontaneous EEG in humans given sub-anaesthetic doses of ketamine. bioRXiv 2019 508697; doi: https://doi.org/10.1101/508697
- [Background] Messner M, Beese U, Romstock J, Dinkel M, Tschaikowsky K. The bispectral index declines during neuromuscular block in fully awake persons. Anesth Analg. 2003 Aug;97(2):488-491. doi: 10.1213/01.ANE.0000072741.78244.C0. PMID 12873942
- [Background] Egerhazi A, Berecz R, Bartok E, Degrell I. Automated Neuropsychological Test Battery (CANTAB) in mild cognitive impairment and in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Apr 13;31(3):746-51. doi: 10.1016/j.pnpbp.2007.01.011. Epub 2007 Jan 16. PMID 17289240
- [Background] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Background] Masuda T, Yamada H, Takada K, Sagata Y, Yamaguchi M, Tomiyama Y, Oshita S. [Bispectral index monitoring is useful to reduce total amount of propofol and to obtain immediate recovery after propofol anesthesia]. Masui. 2002 Apr;51(4):394-9. Japanese. PMID 11995347
- [Background] Struys MM, De Smet T, Versichelen LF, Van De Velde S, Van den Broecke R, Mortier EP. Comparison of closed-loop controlled administration of propofol using Bispectral Index as the controlled variable versus "standard practice" controlled administration. Anesthesiology. 2001 Jul;95(1):6-17. doi: 10.1097/00000542-200107000-00007. PMID 11465585
- [Background] Tufano R, Palomba R, Lambiase G, Giurleo LG. [The utility of bispectral index monitoring in general anesthesia]. Minerva Anestesiol. 2000 May;66(5):389-93. Italian. PMID 10965722
- [Background] Sandin RH, Enlund G, Samuelsson P, Lennmarken C. Awareness during anaesthesia: a prospective case study. Lancet. 2000 Feb 26;355(9205):707-11. doi: 10.1016/S0140-6736(99)11010-9. PMID 10703802
- [Background] Sebel PS, Bowdle TA, Ghoneim MM, Rampil IJ, Padilla RE, Gan TJ, Domino KB. The incidence of awareness during anesthesia: a multicenter United States study. Anesth Analg. 2004 Sep;99(3):833-839. doi: 10.1213/01.ANE.0000130261.90896.6C. PMID 15333419
- [Background] Orser BA, Mazer CD, Baker AJ. Awareness during anesthesia. CMAJ. 2008 Jan 15;178(2):185-8. doi: 10.1503/cmaj.071761. Epub 2007 Dec 11. No abstract available. PMID 18073268
- [Background] Pollard RJ, Coyle JP, Gilbert RL, Beck JE. Intraoperative awareness in a regional medical system: a review of 3 years' data. Anesthesiology. 2007 Feb;106(2):269-74. doi: 10.1097/00000542-200702000-00014. PMID 17264720
- [Background] Errando CL, Sigl JC, Robles M, Calabuig E, Garcia J, Arocas F, Higueras R, Del Rosario E, Lopez D, Peiro CM, Soriano JL, Chaves S, Gil F, Garcia-Aguado R. Awareness with recall during general anaesthesia: a prospective observational evaluation of 4001 patients. Br J Anaesth. 2008 Aug;101(2):178-85. doi: 10.1093/bja/aen144. Epub 2008 May 30. PMID 18515816
- [Background] Xu L, Wu AS, Yue Y. The incidence of intra-operative awareness during general anesthesia in China: a multi-center observational study. Acta Anaesthesiol Scand. 2009 Aug;53(7):873-82. doi: 10.1111/j.1399-6576.2009.02016.x. Epub 2009 Jun 3. PMID 19496761
- [Background] Lewis SR, Pritchard MW, Fawcett LJ, Punjasawadwong Y. Bispectral index for improving intraoperative awareness and early postoperative recovery in adults. Cochrane Database Syst Rev. 2019 Sep 26;9(9):CD003843. doi: 10.1002/14651858.CD003843.pub4. PMID 31557307

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04529304/Prot_000.pdf
  • Informed Consent Form (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT04529304/ICF_002.pdf